CLINICAL TRIAL: NCT05287451
Title: Risk Reducing Salpingectomy With Delayed Oophorectomy as an Alternative to Risk- Reducing Salpingo-oophorectomy in High Risk-Women to Assess the Safety of Prevention - US Cohort Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-1089; NCI-2022-01291 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2022-02-07; First posted 2022-03-18 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Risk-Reducing Salpingectomy-RRS (Other): Can help to lower the risk of ovarian cancer with a delayed removal of 1.
  Interventions: Other: RIsk-Reducing Salpingectomy (RRS)
- Risk-Reducing Oophorectomy-RRO (Other): Can help to lower the risk of ovarian cancer removing both fallopian tubes.
  Interventions: Other: Risk-Reducing Oophorectomy-RRO
- Risk-Reducing Salpingo-Oophorectomy-RRSO (Other): Can help to lower the risk of ovarian cancer as well as the standard-of-care risk-reducing procedure involving the removal of the fallopian tubes and ovaries (risk-reducing salpingo-oophorectomy-RRSO)
  Interventions: Other: Risk-Reducing Salpingo-Oophorectomy-RRSO

INTERVENTIONS:
Other: RIsk-Reducing Salpingectomy (RRS) — complete questionnaires, standard-of-care laparoscopy to check the abdominal area before the assigned procedure
  Arms: Risk-Reducing Salpingectomy-RRS
Other: Risk-Reducing Oophorectomy-RRO — complete questionnaires, standard-of-care laparoscopy to check the abdominal area before the assigned procedure
  Arms: Risk-Reducing Oophorectomy-RRO
Other: Risk-Reducing Salpingo-Oophorectomy-RRSO — complete questionnaires, standard-of-care laparoscopy to check the abdominal area before the assigned procedure
  Arms: Risk-Reducing Salpingo-Oophorectomy-RRSO

SUMMARY:
This is a prospective preference study that will evaluate non-inferiority of the innovative treatment (RRS with delayed RRO) as compared to the standard treatment (RRSO) with respect to high grade serous (ovarian) cancer incidence

DETAILED DESCRIPTION:
The aim of the project is to evaluate RRS with delayed RRO as an alternative for RRSO in BRCA1/2 gene germline mutation carriers with respect to ovarian cancer incidence. We hypothesize that postponement of oophorectomy and consequent menopause to the age of 40-45 (BRCA1) or 45-50 (BRCA2) compared to current standard RRSO at age 35-40 (BRCA1) or 40-45 (BRCA2) will not lead to a significant increase in ovarian cancer risk.

PRIMARY OBJECTIVE:

To evaluate non-inferiority of the innovative treatment (RRS with delayed RRO) as compared to the standard treatment (RRSO) with respect to high grade serous (ovarian) cancer incidence in BRCA1/2 gene germline mutation carriers.

SECONDARY OBJECTIVE:

Incidence of (pre)malignant findings in tubes/ovaries, perioperative morbidity and mortality, incidence of non-ovarian pelvic cancer, breast cancer, prophylactic breast surgery and uptake of risk reducing oophorectomy.

EXPLORATORY OBJECTIVE:

Estimate high grade serous (ovarian) cancer incidence for innovative and standard treatments in BRIP1, RAD51C, and RAD51D gene germline mutation carriers

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Premenopausal women with a documented deleterious mutation in BRCA1, BRCA2, BRIP1, RAD51C, PALB2 and/or RAD51D gene germline mutation.
2. Age 25-40 years for BRCA1 mutation carriers, 25-45 years for BRCA2 and 30-50 years for BRIP1, RAD51C, RAD51D, and PALB2
3. No longer requires fallopian tubes for natural childbearing. Future plans for IVF are acceptable
4. Presence of at least one fallopian tube
5. Participants may have a personal history of non-ovarian malignancy
6. Informed consent must be obtained and documented.

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Postmenopausal status (natural menopause or due to (cancer) treatment)
2. Wish for second stage RRO within two years after RRS (if clear at enrollment)
3. Legally incapable
4. Prior bilateral salpingectomy
5. A personal history of ovarian, fallopian tube, or peritoneal cancer
6. Current clinicals signs, diagnosis, or treatment for malignant disease. Aromatase Inhibitors, Tamoxifen, and Selective Estrogen Receptor Modulators (SERM) are allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 100 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
To evaluate the non-inferiority of the innovative treatment (RRS with delayed RRO) as compared to the standard treatment (RRSO) with respect to high grade serous (ovarian) cancer incidence in BRCA1/2 gene germline mutation carriers. | through study completion, an average of 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Roni Wilke, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (9):
- United States (9):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - WU St Louis, St Louis, Missouri
  - Mount Sinai Health System, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lyndon Baines Johnson General, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org